CLINICAL TRIAL: NCT05008315
Title: Effects of Soft Tissue Mobilization on Postsurgical Adhesions, Pain, Lumbopelvic Muscle Functions, Spinal Mobility, and Posture in Postpartum Women With Caesarean Section
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical trial has been suspended due to a lack of funding
Sponsor: YI-JU TSAI (Other)
Responsible Party: Sponsor-Investigator, YI-JU TSAI, professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKU_adhesion
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Postsurgical Adhesion
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- deep and superficial tissue mobilization group (Experimental): include deep and superficial tissue mobilization
  Interventions: Other: Myofascial abdominal diaphragm release; Other: Direct focused scar release technique; Other: Direct manipulations to visceral structures; Other: pelvic anatomy education
- superficial tissue mobilization group (Active Comparator): superficial tissue mobilization
  Interventions: Other: Myofascial abdominal diaphragm release; Other: Direct focused scar release technique
- control group (Placebo Comparator): Sham (very light hand touch on the same location as the other two groups but without any treatment intention)
  Interventions: Other: pelvic anatomy education; Other: sham
- vaginal delivery group (Other): education session
  Interventions: Other: pelvic anatomy education

INTERVENTIONS:
Other: Myofascial abdominal diaphragm release — Myofascial abdominal diaphragm release
  Arms: deep and superficial tissue mobilization group; superficial tissue mobilization group
Other: Direct focused scar release technique — Direct focused scar release technique
  Arms: deep and superficial tissue mobilization group; superficial tissue mobilization group
Other: Direct manipulations to visceral structures — Direct manipulations to visceral structures
  Arms: deep and superficial tissue mobilization group
Other: pelvic anatomy education — pelvic anatomy education
  Arms: control group; deep and superficial tissue mobilization group; vaginal delivery group
Other: sham — sham
  Arms: control group

SUMMARY:
Postpartum women with C-section receiving deep and superficial tissue mobilization would have better improvement on pain, lumbopelvic muscle functions, spinal mobility, and posture compare to the superficial tissue mobilization and control group

ELIGIBILITY:
vaginal delivery

Inclusion Criteria:

* Natural birth without C-section scar
* Postpartum more than 6 months
* Without any pain in the lumbopelvic region

C-section

Inclusion Criteria:

* Healed C-section scar > six months
* Scar with or without pain

Both mode of delivery

Exclusion Criteria:

* Active infection or infectious disease in the pelvis or abdomen
* Pain medications on days of measurements
* Skin irritation and inflammation at the site of the scar
* Currently pregnant or actively trying to get pregnant
* History of radiation to the area
* Any fracture around spine and pelvis
* Any previous gynecologic and obstetric surgery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Scar Characteristic: Extensibility | 8 weeks
  The extensibility of the scar will be measured using the modified adheremeter in each of 4 directions including superior, inferior, medial and lateral and then the area of mobility will be calculated.
Scar Characteristic: Viscoelasticity | 8 weeks
  The biomechanical and viscoelastic properties of the scar tissue will be measured using a non-invasive myometer
Scar Characteristic: Irritability | 8 weeks
  The irritability of the scar will be measured using the digital pressure algometer for two conditions: first, when the pressure turns from discomfort to pain and the participant asks to stop, and then when the maximal pressure or pain the participant can tolerate.
Muscle function measures of lumbopelvic muscles | 8 weeks
  Ultrasonography image for muscle thickness of lumbopelvic muscles during rest and maximum contraction.
Muscle function measures of pelvic floor muscle control | 8 weeks
  Ultrasonography image for muscle thickness of pelvic floor muscle control during rest, maximum contraction
Spinal Mobility | 8 weeks
  Range of motion for cervical, thoracic, and lumbar spine in the sagittal, frontal, and transverse plane as well as pelvic tilt will be assessed using the wireless double inclinometers
Myofascial Flexibility | 8 weeks
  Straight leg raise test and Thomas test will be used to examine the muscle flexibility of the major lower extremity muscles.
Spinal Alignment and Posture | 8 weeks
  Radiographic measurement, posture will be assessed using the photographic measurement. Reflective markers will first be placed and attached on the canthus of the eye, tragus of the ear, the spinous processes of C2, C7, T1, T3, T11, T12, L1, L5, S1, S5, and bilateral anterior superior iliac spine and posterior superior iliac spine in standing. The participants will be instructed to maintain their gaze straight ahead at a target adjusted for body height. Two standing photographs will be taken, one in the usual standing posture and the other in the best standing posture. Following the other two photographs will be taken, one in maximal pelvic anterior tilt and the other in the maximal pelvic posterior tilt.
Pain intensity measure of Visual Analogue Scale | 8 weeks
  Visual Analogue Scale is a self-reported instrument assessing average pain intensity in currently. Possible score range from 0 (no pain) to 10 (worst possible pain).
Pain intensity measure of pelvic girdle questionnaire | 8 weeks
  pelvic girdle questionnaire is a self-reported instrument assessing pelvic girdle pain intensity in currently. Questionnaire consisting of 20 activity items and 5 symptom items on a 4-point response scale. Possible score range from 0 (no pain) to 100 (worst possible pain).
Pain intensity measure of Oswestry Low Back Pain Disability Questionnaire | 8 weeks
  Oswestry Low Back Pain Disability Questionnaire is a self-reported instrument assessing patient's permanent functional disability in currently. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. The higher the score, the greater the degree of disability.

SECONDARY OUTCOMES:
Self-perceived Change Health Status: Global Rating of Change Scale (GROC) | 8 weeks
  The GROC is a single-item instrument that provides a means of measuring self-perceived change in health status. The GROC uses the 15-point Likert scale to rate the perceived "overall change" on a continuum, with -7 (labeled "worse") on the left and +7 (labeled "better") on the right, and 0 in the middle (labeled "no change"), compared with the baseline
Patient and Observer Scar Assessment Scale (POSAS) | 8 weeks
  The POSAS includes 2 numerical numeric scales: The Patient Scar Assessment Scale and the Observer Scar Assessment Scale. It objectively assesses vascularity, pigmentation, thickness, relief, pliability, and surface area, and incorporates patient subjective symptoms of pain, itching, color, stiffness, thickness, and relief.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Tainan, Taiwan